CLINICAL TRIAL: NCT04372563
Title: Clinical Study of Diagnosis and Treatment of Thoracic Aortic Aneurysms and Dilatation in Combination With Tricuspid and Bicuspid Aortic Valves.
Brief Title: Study of Treatment of Thoracic Aortic Aneurysms and Dilatation in Combination With Tricuspid and Bicuspid Aortic Valves.
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Evgenia V. Lelik, researcher, Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: Aortic Aneurysm & Dilation
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Ascending Aorta Aneurysm; Dilation of the Ascending Aorta
MeSH Terms: conditions — Aneurysm, Ascending Aorta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy: Healthy patients with normal aortic dimensions
  Interventions: Other: aortic prosthetics
- ascending aortic dilation 45-55, operated on: patients with ascending aortic dilation 45-55, tricuspid aortic valves operated on
  Interventions: Other: aortic prosthetics
- ascending aortic dilation 45-55, non operated on: patients with ascending aortic dilation 45-55, tricuspid aortic valves non operated
  Interventions: Other: aortic prosthetics

INTERVENTIONS:
Other: aortic prosthetics — aortic prosthetics

SUMMARY:
Clarification of indications for surgical correction in patients with borderline expansion of the ascending aorta

DETAILED DESCRIPTION:
Expanding indications for surgical treatment of patients with borderline values of the ascending aorta

ELIGIBILITY:
Inclusion Criteria:

1. Extension of the ascending aorta less than 55 mm
2. Tricuspid Aortic Valves.
3. Extension of the ascending aorta more than 45 mm

Exclusion Criteria:

1. Age less 45 years
2. Age more 75 years
3. Multiple organ failure
4. oncological disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with computed tomography-diagnosed ascending aortic dilation greater than 45 mm, less than 55 mm with tricuspid aortic valve compared to patients with bicuspid aortic valve and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
death | 30 day after operation
  death
aorto-associated complications | 30 day
  rupture, dissection

SECONDARY OUTCOMES:
increasing the diameter of the ascending aorta | 1 year
  increasing the diameter of the ascending aorta more than 55 mm

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniya V Lelik, PhD, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (2):
- Russia (2):
  - Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk
  - Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk

IPD SHARING:
Plan to Share IPD: No